CLINICAL TRIAL: NCT05767736
Title: An Observational Study Utilising Data From Big MS Data Registries to Evaluate the Long-Term Safety of Vumerity and Tecfidera
Brief Title: A Study to Evaluate Long-Term Safety of Vumerity and Tecfidera in Participants With Multiple Sclerosis (MS)
Status: Active, not recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 272MS403; EUPAS1000000285 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — diroximel fumarate; Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Vumerity Cohort: Participants who have been prescribed Vumerity as a newly initiating treatment and not previously treated with Tecfidera are selected and the available data is collected retrospectively.
  Interventions: Drug: Diroximel Fumarate
- Tecfidera Cohort: Participants who have been prescribed Tecfidera as a newly initiating treatment and not previously treated with Vumerity are selected and the available data is collected retrospectively.
  Interventions: Drug: Dimethyl Fumarate
- Vumerity/Tecfidera Switch Cohort: Participants who have been treated with Tecfidera and then switched to Vumerity as per routine medical care are selected and the available data is collected retrospectively.
  Interventions: Drug: Diroximel Fumarate; Drug: Dimethyl Fumarate
- Selected Disease Modifying Therapies (DMTs) Treated Cohort: Participants who have been prescribed with other selected DMTs (teriflunomide, beta-interferons, or glatiramer acetate) and are not previously treated with Vumerity or Tecfidera are selected and the available data is collected retrospectively.
  Interventions: Drug: Disease-Modifying Therapies (DMTs)

INTERVENTIONS:
Drug: Diroximel Fumarate — Administered as specified in the treatment arm.
  Other Names: VUMERITY; BIIB098
  Groups: Vumerity Cohort; Vumerity/Tecfidera Switch Cohort
Drug: Dimethyl Fumarate — Administered as specified in the treatment arm.
  Other Names: Tecfidera; DMF; BG00012
  Groups: Tecfidera Cohort; Vumerity/Tecfidera Switch Cohort
Drug: Disease-Modifying Therapies (DMTs) — Administered as specified in the treatment arm.
  Groups: Selected Disease Modifying Therapies (DMTs) Treated Cohort

SUMMARY:
The primary objective of the study is to estimate the incidence rate of serious adverse events (SAEs), including but not limited to malignancies and serious and opportunistic infections, among participants with MS treated with Vumerity, Tecfidera, other selected disease modifying therapies (DMTs [teriflunomide, beta interferons, or glatiramer acetate]), or Vumerity after switching from Tecfidera. The secondary objective of the study is to compare the incidence rate of SAEs, including but not limited to malignancies and serious and opportunistic infections, among MS participants treated with Vumerity, Tecfidera, and Vumerity after switching from Tecfidera with the incidence rate of MS participants treated with other selected DMTs (teriflunomide, beta-interferons, or glatiramer acetate), if the sample size allows.

ELIGIBILITY:
Key Inclusion Criteria:

- Participants with MS treated with at least 1 dose of Vumerity, Tecfidera, or other selected DMTs (teriflunomide, beta-interferons, or glatiramer acetate), and whose data are captured in the BMSD network will be included in the study.

Key Exclusion Criteria:

- None

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with MS who are treated with Vumerity, Tecfidera, or other selected DMTs (teriflunomide, beta-interferons, or glatiramer acetate) at the initiation of the treatment and participating in Big Multiple Sclerosis Data (BMSD) network registry.
Sampling Method: Probability Sample
Enrollment: 10500 (Estimated)
Dates: Start 2024-06-08 (Actual); Primary Completion 2032-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Confirmed Serious Adverse Events (SAEs) in the Vumerity, Tecfidera, Other Selected DMTs (Teriflunomide, Beta-interferons, or Glatiramer Acetate), or Vumerity/Tecfidera Switch Cohorts | Up to 10 years
  An SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, and results in a congenital anomaly/birth defect. The incidence rate of confirmed SAEs, will include but not be limited to malignancies and serious and opportunistic infections among participants with MS who are treated with Vumerity, Tecfidera, and other selected DMTs (teriflunomide, beta-interferons, or glatiramer acetate).

SECONDARY OUTCOMES:
Hazard Ratio of Confirmed SAEs in Vumerity, Tecfidera, or Vumerity/Tecfidera Switch Cohorts Versus Other Selected DMTs (Teriflunomide, Beta-interferons, or Glatiramer acetate) Cohort | Up to 10 years
  An SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, and results in a congenital anomaly/birth defect. The incidence rate of confirmed SAEs, will include but not be limited to malignancies and serious and opportunistic infections among participants with MS who are treated with Vumerity, Tecfidera, or other selected DMTs (teriflunomide, beta-interferons, or glatiramer acetate).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org